CLINICAL TRIAL: NCT02795572
Title: Protocol Comparing a Nutraceutical Formulation Consisting of Omega-3 Fatty Acids, Vitamin D, and Vitamins B6 Plus B12 Versus No Treatment in the Prevention or Reduction of Chemotherapy Induced Peripheral Neuropathy (CIPN) in Patients Treated With Docetaxel as Neoadjuvant/Adjuvant Breast Cancer Therapy
Brief Title: Nutraceuticals Versus Usual Care in the Prevention or Reduction of CIPN in Patients Treated With Docetaxel as Neoadjuvant/Adjuvant Breast Cancer Therapy
Acronym: CIPN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Retirement of the Principal Investigator
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIPNN-SMG-CCI-01
Record Dates: First submitted 2016-05-30; First posted 2016-06-10 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Peripheral Neuropathy in Breast Cancer Patient
Keywords: Breast Neoplasms; Peripheral Neuropathies
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases | interventions — Vitamin D; Vitamin B 6; Vitamin B 12; Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive a daily dose of Vitamin D 2000 IU, Vitamin B6 100 mg, Vitamin B12 100 mcg and Omega-3 Fatty Acids 2700 mg [900 mg TID (600 mg EPA, 300 mg DHA)].
  Interventions: Dietary Supplement: Vitamin D; Dietary Supplement: Vitamin B6; Dietary Supplement: Vitamin B12; Dietary Supplement: Omega-3 Fatty Acids
- Reference Group (No Intervention): Reference group will receive usual care.

INTERVENTIONS:
Dietary Supplement: Vitamin D — Vitamin D 2000 IU oral once daily
  Arms: Intervention Group
Dietary Supplement: Vitamin B6 — Vitamin B6 100 mg oral once daily
  Arms: Intervention Group
Dietary Supplement: Vitamin B12 — Vitamin B12 100 mcg oral once daily
  Arms: Intervention Group
Dietary Supplement: Omega-3 Fatty Acids — Omega-3 Fatty Acids 900 mg oral three times a day (600 mg EPA, 300 mg DHA)
  Arms: Intervention Group

SUMMARY:
The trial will utilize Nutraceuticals (Vitamin D 2000IU oral once daily, Vitamin B6 100 mg oral once daily, Vitamin B12 100 mcg oral once daily, Omega-3 Fatty Acids 900 mg oral three times a day) in patients treated with Docetacel as Neoadjuvant or Adjuvant Breast cancer Therapy. The trial is being conducted to see if the use of Nutraceuticals will prevent or reduce Chemotherapy Induced Peripheral Neuropathy (CIPN).

DETAILED DESCRIPTION:
Phase 2, Single Centre, Open-label 2 Arm Randomized Trial. The intervention group will receive a daily dose of Vitamin D, Omega-3-fatty acids, Vitamin B6, and Vitamin B12. The reference group will have usual care.

Dose of Nutraceuticals: Vitamin D 2000 IU oral once daily, Vitamin B6 100 mg oral once daily, Vitamin B12 100 mcg oral once daily, Omega-3 Fatty Acids 900 mg oral three times a day (600 mg EPA, 300 mg DHA)

Population: Breast Cancer patients undergoing either neoadjuvant or adjuvant therapy with docetaxel.

106 participants in total will be needed with accrual being completed in hopefully 1 years' time. Study Investigators will screen the candidates for the study.

ELIGIBILITY:
Inclusion Criteria:

* Female 18-70 years of age
* Biopsy proven invasive breast carcinoma
* Scheduled to receive docetaxel (3-6 cycles)
* Have values for liver (AST, ALT, Bilirubin) and renal function (CREAT), within 1.5 times normal values as drawn per standard of care.
* ECOG 0-2
* Be able to provide informed consent
* Willingness to adhere to regimen

Exclusion Criteria:

* Metastatic disease
* Any peripheral neuropathy
* Known HIV (testing not required)
* Diseases causing malabsorption i.e.: Inflammatory Bowel Disease, Celiac and Whipple's Disease
* Patients with seafood allergies
* Patients on Warfarin or with a documented clinically significant bleeding disorder

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Chemotherapy Induced Peripheral Neuropathy Assessment | 12 months
  To determine if there is a reduction in either severity or incidence of CIPN in patients treated with docetaxel in the female breast cancer population by using a nutraceutical formulation of the investigators design.

SECONDARY OUTCOMES:
Delay in the onset of grade 1 or decrease in the severity of CIPN | 12 months after initiation of chemotherapy
Affect of Usage of Nutraceuticals on Response to treatment | 24 months

OTHER OUTCOMES:
Association of specific SNPs to CIPN | 24 months
Association of SNPs and Therapeutic response | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Katia Tonkin, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No